CLINICAL TRIAL: NCT05097313
Title: Evaluation of the Antioxidant and Immunomodulatory Effect of a β-glucan Fiber From Saccharomyces Cerevisiae in Healthy Adults, Medellín - Antioquia 2021-2022
Brief Title: Antioxidant and Immunomodulatory Effect of a β-glucan Fiber From Saccharomyces Cerevisiae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Levapan S.A (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PEC02_2020
Record Dates: First submitted 2021-08-27; First posted 2021-10-28 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Nutrition, Healthy
Keywords: B-glucan; Saccharomyces cerevisiae; Antioxidant; Inmunomodulador

STUDY DESIGN:
Intervention Model Description: This is an interventional, randomized, non-comparative, exploratory, three-arm, double-blind, randomized study, divided into three groups (2 intervention and placebo) using an allocation ratio of 1: 1: 1.
  Treatment allocation will be made according to a random code.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind trial. Research product blinding will be maintained using one label for both products (fiber and placebo) and the same capsules for both.
  Subjects, who collect the data (eg, Investigator and coordinator) and those who evaluate the data (eg, Statistician) will be blinded. One or more pharmacists / vaccine administrators designated by the facility will not be blinded. These designated unblinded individuals will maintain investigational vaccine blindness and will not participate in the safety assessment of the subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- consumption of 250 mg of β-glucan (Experimental): Patients with oral consumption of 250 mg (one capsule) of β-glucan from Yeast Plus once a day for 84 days without interruption.
  Interventions: Dietary Supplement: Yeast β-glucan fiber
- consumption of 500 mg of β-glucan (Experimental): Patients with oral consumption of 500 mg (two capsules) of β-glucan from Yeast Plus once a day for 84 days without interruption.
  Interventions: Dietary Supplement: Yeast β-glucan fiber
- 200 mg or 400 mg placebo (Placebo Comparator): Placebo patients, with oral soy protein consumption, half of the group 200 mg (one capsule) and the remaining 400 mg (two capsules) once a day for 84 days without interruption
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Yeast β-glucan fiber — The study is designed to determine if β-glucan is safe and if it presents an antioxidant and immunomodulatory response in healthy adults in Colombia.
  Other Names: β-glucan
  Arms: consumption of 250 mg of β-glucan; consumption of 500 mg of β-glucan
Other: Placebo — oral consumption of 200 mg (one capsule) or 400 mg (two capsules) of soy protein powder for 84 days.
  Arms: 200 mg or 400 mg placebo

SUMMARY:
Β-glucans are linear polymers of glucose of high molecular weight that are found naturally in the cell wall of various living organisms such as bacteria, yeast, fungi and plants; They are widely used in food companies as texturizers.

Scientific studies suggest that the consumption of β-glucans would be associated with benefits for human health such as reducing the risk of cardiovascular diseases and strengthening the immune system. These effects depend on their source of origin; those from cereals have been attributed beneficial metabolic properties and those that come from yeast immunostimulating properties.

Yeast β-glucans are believed to be potent immunomodulators with effects on innate and adaptive immunity. This effect could be due to the ability to stimulate receptors of the immune system present in the membrane of enterocytes, M cells and dendritic cells, improving the phagocytic activity of macrophages and the antimicrobial activity of mononuclear cells and neutrophils.

Due to this property, β-glucans are being used more and more for the development of functional foods in several countries of the world. However, the effect of yeast β-glucans on the stimulation of the immune response has not yet been accurately documented; Therefore, the present investigation aims to establish the performance of a β-glucan fiber from S. cerevisiae in antioxidant and immunomodulatory activity in healthy volunteers.

DETAILED DESCRIPTION:
Background

Β-glucans are high molecular weight glucose polymers (polysaccharides) naturally present in the cell wall of various living organisms such as bacteria, yeast, fungi and plants. Some studies show that β-glucans have antioxidant activity and stimulate the immune system in animals and humans.

On the other hand, the physiological metabolism in living beings generates free radicals that can endanger cell integrity if they are not controlled properly. Free radicals are collectively known as Reactive Oxygen Species (ROS) and have the ability to produce significant oxidative damage to cellular structures that can increase under environmental stress. Free radicals impair tissue function, contribute to aging and the development of chronic and chronic degenerative diseases.

To counteract the action of free radicals, antioxidants are used whose function is to maintain or restore cellular balance. An alternative for this are β-glucans since they have protective properties against oxidative damage, the antioxidant effect they exert is indirect and is produced by improving the expression and production of antioxidant systems by the body itself.

Various studies focused on antioxidant activity indicate that β-glucans from mushrooms constitute a potential natural source of antioxidants, especially associated with regular consumption.

Added to the effects caused by ROS is the constant exposure of living beings to pathogens, which must be dealt with by the immune system through cells and tissues to avoid infections. The immune system, made up of the innate and the adaptive systems, is essential for survival as it protects the body against potentially dangerous microorganisms that constantly attack the human body. Therefore, the proper functioning of the immune system must be guaranteed, since limitations in it increase the possibility of contracting serious infections that threaten life. In accordance with this, it is reported that changes in dietary composition can improve immune function. Although studies have been reported in the literature since 1939 on the response of the immune system by yeast cell walls, it is in the 1960s that it is established that the active substance in yeast that generates the beneficial effect is β -glucan. Β-glucans are known as biological response modifiers, due to their ability to activate the immune system, since they favor the participation of immune cells in a greater proportion in the face of external threats.

In the same way, the scientific literature indicates that there are various properties attributed to the use of β-glucan, among them the decrease in allergy episodes, respiratory tract infections, decreased concentrations of glycoproteins of the immune system and increased potential of blood leukocytes to produce IL-2, IL-4, IL-5, and interferon (IFN-γ), the foregoing, suggesting that β-glucans hold promise for modulating an individual's immunity .

In this sense, the company Levapan SA multilatina company of Colombian origin founded in 1953, which is dedicated to the production and commercialization of yeast (S. cerevisiae), yeast extracts, flavor enhancers, raw materials for food industries, bakery and confectionery, mass consumption products, gastronomy, agribusiness, vegetable and animal proteins, has worked on the production of β-glucan from S. cerevisiae, showing potential effects on health.

Within its portfolio, the product derived from yeast that is currently used as an ingredient in different formulations of the nutraceutical industry is presented as β-glucan Plus, since they offer immunostimulating properties. It is also considered that β-glucan may be a promising alternative to control or mitigate the effects of the SARS-CoV-2 virus responsible for the COVID-19 disease. However, it is necessary to evaluate and confirm the antioxidant and immunomodulatory effect of β-glucan Plus through a clinical evaluation as proposed by this research.

Benefits of β-glucan

Evidence supports that the inclusion of these polysaccharides in the diet can have positive effects on glycemic control, cholesterol and immunity. Due to their physical and chemical characteristics, they have been used during the development of functional foods to improve their texture and shelf life. Β-glucans are related to anti-inflammatory, antiviral, antioxidant, and immunomodulatory activity. Antimutagenic, chemoprotective and anticancer effects of these compounds have also been reported and they are reported to have positive effects on cardiovascular diseases, arteriosclerosis, diabetes, wound healing.

Currently, β-glucan extracted from microorganisms is being used for the treatment of many diseases in the world. Processes have been carried out to extract β-glucans from the cell wall of S. cerevicie and develop products with it. However, work continues to obtain evidence to demonstrate its effectiveness through clinical studies.

Global situation due to the COVID-19 pandemic

The spread of the COVID-19 virus) has prompted interest in boosting immunity. With this perspective Kerry notes that clinical research has shown that his Wellmune β-glucan can help support upper respiratory tract infections. The company says it can support the immune system of people, including children, athletes, older adults and those with lifestyle stress. Wellmune notes that a healthy immune system is the best defense against disease, although there is no specific research demonstrating Wellmune's effectiveness against diseases like COVID-19.

Treatments with β-glucan. At present there is an interest in promoting the immune response of organisms in a natural way, these facts have motivated the interest in conducting research on the immunomodulatory effect derived from natural systems. These scientific studies suggest that its consumption would be associated with benefits for human health such as reducing the risk of cardiovascular diseases and strengthening the immune system. These effects depend on their source of origin, those from cereals have been attributed beneficial metabolic properties and those that come from yeast immunostimulating properties; According to this theory, yeast β-glucans are believed to be potent immunomodulators with effects on innate and adaptive immunity. This effect could be due to the ability to stimulate receptors of the immune system present in the membrane of enterocytes, M cells and dendritic cells, improving the phagocytic activity of macrophages and the antimicrobial activity of mononuclear cells and neutrophils.

Β-glucan from bakery yeast produced by Levapan S.A

The β-glucan of Yeast Plus is a product of Levapan SA that contains 1,3 and 1,6 Β- Glucan extracted under hydrolysis processes of the cell wall of the yeast S. cerevisiae, where at the end of the process a product is obtained insoluble in water. The product is originated from non-genetically modified microorganisms, baker's yeast is the primary yeast made from sugar cane molasses. Annually the company produces approximately 20 Ton / month of β-glucan for its use in different formulations, such as the development of nutraceutical foods for human consumption, animal feed, aquaculture, among others.

The β-glucan Plus is currently manufactured by Levapan S. A company that has the KOSHER, HALAL and ISO 9001: 2008 certifications for the production and preparation of glucan and is evaluated by PECET following the BPC protocols.

There are extensive properties attributable to β-glucans that allow evaluating their actions in various fields, being used more and more for the development of functional foods in various countries of the world, but with few results that demonstrate the real effect of these.

Due to these properties there are several studies focused on the effects of β-glucans, however, the effect of β-glucans from yeast S. cerevisiae on the stimulation of the immune response has not yet been accurately documented, so the This research aims to establish the performance of a S. cerevisiae β-glucan fiber in antioxidant and immunomodulatory activity in healthy volunteers.

Due to the antioxidant and immunomodulatory activity of the different types of β-glucans, these are being used more and more for the development of functional foods in several countries of the world. However, the effect of yeast β-glucans on the stimulation of the immune response has not yet been accurately documented; Therefore, the present investigation aims to establish the performance of a β-glucan fiber from S. cerevisiae in antioxidant and immunomodulatory activity in healthy volunteers.

OBJECTIVES OF THE STUDY

General objective

To determine the antioxidant and immunomodulatory effect of a β-glucan fiber obtained from the yeast S. cerevisiae in healthy adults.

Specific objectives

* Determine the antioxidant activity of a β-glucan fiber obtained from S.cerevisiae
* To determine the strengthening of the immune system of a β-glucan fiber obtained from the yeast S. cerevisiae
* Evaluate the safety and tolerability (frequency, seriousness and degree of adverse events) of a β-glucan fiber obtained from the yeast S. cerevisiae
* Explore the metabolic benefit of a β-glucan fiber obtained from the yeast S. cerevisiae
* Explore the impact of the consumption of a β-glucan fiber obtained from the yeast S. cerevisiae on the severity of the SARS-CoV-2 coronavirus infection

ELIGIBILITY:
Inclusion criteria

* Men and women aged ≥18 and ≤45 years without abnormal findings at the time of physical examination
* Tests of creatinine, transaminases, lipid profile, glycemia and hemogram with ranges of normality according to laboratory reference values and / or at the discretion of the researcher
* Body Mass Index (BMI) between 18.5 and 25 kg / m2
* In the opinion of the researcher, the participant is able to understand and comply with the protocol

Exclusion criteria

* Women with a positive pregnancy test during the screening process or who do not agree with the use of a contraceptive method until day 90 post-treatment
* Women who are breastfeeding
* Clinically significant pathological history such as kidney disease, hypertension, diabetes, anemia, autoimmune or psychiatric diseases, among others that may affect the development or results of the study.
* Manifest eating styles other than the omnivore
* Have food restrictions derived from allergic, metabolic, dermatological diseases, lithiasis, irritable bowel and / or health conditions that imply permanent modification in diet
* Consumption of a vitamin or nutritional supplement
* Any condition that, in the opinion of the investigator, may affect the development of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Antioxidant capacity | Day 140
  Evaluation of antioxidant capacity of β-glucan Fiber through analysis of results of tests from Baseline level compared to day 42, day 84 and day 140.
Immunomodulatory capacity | Day 140
  Evaluation of immunomodulatory capacity of β-glucan Fiber through analysis of results of tests from Baseline level compared to day 42, day 84 and day 140.

SECONDARY OUTCOMES:
Metabolic benefit | Day 140
  Changes of lipid profile in participants. Changes from Baseline level compared to day 42, day 84 and day 140 evaluations
Metabolid benefit | Day 140
  Changes of glucose level in participants. Changes from Baseline level compared to day 42, day 84 and day 140 evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Iván D Vélez, MD. PhD., Principal Investigator — Director PECET
Locations (1):
- Program for Research and Control in Tropical Diseases - PECET, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Corno M, Gessani S, Conti L. Shaping the Innate Immune Response by Dietary Glucans: Any Role in the Control of Cancer? Cancers (Basel). 2020 Jan 8;12(1):155. doi: 10.3390/cancers12010155. PMID 31936360
- [Background] Pérez-Guisado J. Arguments in favor of incorporating β-D-glucans in food. Endocrinología y Nutrición. 2007;54(6):315-24.
- [Background] Divya M, Gopi N, Iswarya A, Govindarajan M, Alharbi NS, Kadaikunnan S, Khaled JM, Almanaa TN, Vaseeharan B. beta-glucan extracted from eukaryotic single-celled microorganism Saccharomyces cerevisiae: Dietary supplementation and enhanced ammonia stress tolerance on Oreochromis mossambicus. Microb Pathog. 2020 Feb;139:103917. doi: 10.1016/j.micpath.2019.103917. Epub 2019 Dec 10. PMID 31830581
- [Background] Antioxidant Effect of Beta-glucan Extract from Saccharomyces Cerevisiae. Indian Journal of Forensic Medicine & Toxicology. 2020.
- [Background] Vetvicka V, Vannucci L, Sima P, Richter J. Beta Glucan: Supplement or Drug? From Laboratory to Clinical Trials. Molecules. 2019 Mar 30;24(7):1251. doi: 10.3390/molecules24071251. PMID 30935016
- [Background] Carvajal Carvajal C. Reactive oxygen species: formation, function and oxidative stress. Legal Medicine of Costa Rica. 2019; 36: 91-100.
- [Background] Özcan Ö, Ertan F. Beta-glucan Content, Antioxidant and Antimicrobial Activities of Some Edible Mushroom Species. Food Science and Technology. 2018;6(2):47-55.
- [Background] Zrnic-Ciric M, Dabetic N, Todorovic V, Djuris J, Vidovic B. Beta-glucan content and antioxidant activities of mushroom-derived food supplements. Journal of the Serbian Chemical Society. 2020;85(4):439-51.
- [Background] Song H-S, Moon K-Y. In vitro antioxidant activity profiles of ${\beta} $-glucans isolated from yeast Saccharomyces cerevisiae and mutant Saccharomyces cerevisiae IS2. Food Science and Biotechnology. 2006;15(3):437-40.
- [Background] Volman JJ, Mensink RP, Ramakers JD, de Winther MP, Carlsen H, Blomhoff R, Buurman WA, Plat J. Dietary (1-->3), (1-->4)-beta-D-glucans from oat activate nuclear factor-kappaB in intestinal leukocytes and enterocytes from mice. Nutr Res. 2010 Jan;30(1):40-8. doi: 10.1016/j.nutres.2009.10.023. PMID 20116659
- [Background] Carpenter KC, Breslin WL, Davidson T, Adams A, McFarlin BK. Baker's yeast beta-glucan supplementation increases monocytes and cytokines post-exercise: implications for infection risk? Br J Nutr. 2013 Feb 14;109(3):478-86. doi: 10.1017/S0007114512001407. Epub 2012 May 10. PMID 22575076
- [Background] Pizarro C S, Ronco M AM, Gotteland R M. ß-glucans: what types are there and what are their health benefits? Chilean nutrition magazine. 2014; 41: 439-46.
- [Background] Talbott SM, Talbott JA, Talbott TL, Dingler E. beta-Glucan supplementation, allergy symptoms, and quality of life in self-described ragweed allergy sufferers. Food Sci Nutr. 2013 Jan;1(1):90-101. doi: 10.1002/fsn3.11. Epub 2014 Jan 8. PMID 24804018
- [Background] Kirmaz C, Bayrak P, Yilmaz O, Yuksel H. Effects of glucan treatment on the Th1/Th2 balance in patients with allergic rhinitis: a double-blind placebo-controlled study. Eur Cytokine Netw. 2005 Jun;16(2):128-34. PMID 15941684
- [Background] Espinoza-Gallardo D, Contreras-Porcia L, Ehrenfeld N. ß-glucans, their production and properties in microalgae with emphasis on the genus Nannochloropsis (Ochrophyta, Eustigmatales). Journal of Marine Biology and Oceanography. 2017; 52 (1): 33-49.
- [Background] San Mauro-Martín I, Garicano Vilar E. Role of vitamin C and β-glucans on the immune system: review. Spanish Journal of Human Nutrition and Dietetics. 2015; 19 (4): 238.
- [Background] Lazaridou A, Biliaderis CG. Molecular aspects of cereal β-glucan functionality: Physical properties, technological applications and physiological effects. J Cereal Sci. 2007;46(2):101-18.
- [Background] Vásquez-Piñeros MA, Rondón-Barragan IS, Eslava-Mocha PR. Immunostimulants in teleost fish: probiotics, B-glucans and lipopolysaccharides. Orinoquia. 2012;16(1):46-62.
- [Background] Brennan CS CL. The potential use of cereal (1→3,1→4)-β-d-glucans as functional food ingredients. J Cereal Sci. 2005;42(1):1-13.
- See also: TERRA HD. Beta-glucans: immune regulators and cardiovascular protectors 2019 — https://hifasdaterra.com/blog/beta-glucanos-reguladores-inmunitarios-y-protectores-cardiovasculares/
- See also: nutritioninsight. Lallemand Bio-Ingredients adquiere Biotec BetaGlucans para expandir la estrategia de levadura beta-glucano 2020 — https://www.nutritioninsight.com/news/lallemand-bio-ingredients-acquires-biotec-betaglucans-to-expand-beta-glucan-yeast-strategy.html